CLINICAL TRIAL: NCT00273481
Title: Cosopt Versus Xalacom
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmaceutical Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRN 05-001
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — dorzolamide; Timolol; Latanoprost

INTERVENTIONS:
Drug: dorzolamide 2%/timolol maleate 0.5% fixed combination
Drug: latanoprost 0.005%/timolol maleate 0.5% fixed combination
Drug: timolol maleate 0.5%
Drug: placebo

SUMMARY:
To compare the intraocular pressure efficacy and safety of the DTFC given twice daily versus the LTFC given once every morning following a run-in period with timolol maleate given twice daily.

ELIGIBILITY:
Inclusion Criteria:

* adults with primary open-angle or pigment-dispersion glaucoma, or ocular hypertension
* at baseline the intraocular pressure should be 20 to 32 mm Hg inclusive at 08:00 measurement (Visit 2) after dosing with timolol the evening before
* the intraocular pressure should be 32 mm Hg or less at all the time points in both eyes at Visit 2
* visual acuity should be 6/60 or better in the study eye(s)

Exclusion Criteria:

* any anticipated change in systemic hypotensive therapy during the trial
* use of any corticosteroids by any route for more than two weeks during the study
* contraindications to study medicines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33
Dates: Start 2005-09; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Stewart, MD, Study Director — Pharmaceutical Research Network, LLC; Cindy M. Hutnik, BSc, PhD, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Barbara Cvenkel, MD, Principal Investigator — University Eye Clinic Ljubljana
Locations (2):
- Lawson Health Research Insitute, London, Ontario, Canada
- University Eye Clinic, Ljubljana, Slovenia